CLINICAL TRIAL: NCT04210128
Title: Continuous Glucose Monitoring For Prediction and Treatment of Steroid-Induced Hyperglycemia
Brief Title: Glucose Monitoring to Predict and Treat High Glucose Levels After Steroid Treatment
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 19-315
Record Dates: First submitted 2019-12-20; First posted 2019-12-24 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer; Pancreatic Cancer; Diabetes; Pre Diabetes
Keywords: Glucose Monitoring; 19-315
MeSH Terms: conditions — Breast Neoplasms; Pancreatic Neoplasms; Diabetes Mellitus; Glucose Intolerance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast cancer patients: A blinded continuous glucose monitor (specifically a Freestyle Libre Pro) will be worn for a 14 day period by patients during the first and third cycles of breast neoadjuvant chemotherapy. At the end of that period (after completion of the one round of chemotherapy) readings will be downloaded from the sensor and the sensor will be removed. Readings will be evaluated by the treating endocrinologist as well as the study team and appropriate clinical interventions.
- Pancreatic cancer patients: A blinded continuous glucose monitor (specifically a Freestyle Libre Pro) will be worn for a 14 day period by patients during the first and third cycles of pancreatic chemotherapy. At the end of that period (after completion of the one round of chemotherapy) readings will be downloaded from the sensor and the sensor will be removed. Readings will be evaluated by the treating endocrinologist as well as the study team and appropriate clinical interventions.

SUMMARY:
The purpose of this study is to see if continuous glucose monitoring can identify how often people who have pre-diabetes or medical obesity or well-controlled diabetes experience very high glucose values while receiving chemotherapy for breast cancer or pancreatic.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or older undergoing neoadjuvant chemotherapy regimens including taxane and/or anthracycline for breast cancer.
* Patient aged 18 or older undergoing any chemotherapy regimen for pancreatic cancer
* Have 'high metabolic risk(either pre-diabetes, obesity, or well-controlled diabetes) defined as either:

  * Pre-diabetes and/or obesity group: one or more of known HbA1c 5.7-6.5%, fasting glucose > 100 mg/dL, or BMI > 30
  * Well-controlled diabetes: Known HbA1c < 7.5 on lifestyle alone or up to one oral antidiabetic agent
  * Any patient undergoing treatment for pancreatic adenocarcinoma on either no antidiabetic agent or up to one oral antidiabetic agent

Exclusion Criteria:

* Patients with type 1 diabetes, a history of hospitalization for either hyperglycemia or ketoacidosis, a history of hypoglycemia requiring hospitalization, rashes or other skin reactions that would preclude placement of the CGM
* Use of anticoagulants or antiplatelet agents other than aspirin
* Platelet count < 50 K/μL within 60 days prior to enrollment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer
Study Population: Patients will be recruited through the breast and gastrointestinal (GI) medicine oncology clinics at MSKCC.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
severe hyperglycemia | 1 year
  glucose > 400 mg/dL for over 3 contiguous hours

CONTACTS AND LOCATIONS:
Overall Officials: James Flory, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm